CLINICAL TRIAL: NCT02723032
Title: Validation of a Miniature SpO2 Sensor in Healthy Subjects and Patients With Long-term Oxygen Therapy. A Prospective, Method Comparison, Proof of Concept Study.
Brief Title: Validation of a Miniature SpO2 Sensor in Healthy Subjects and Patients With Long-term Oxygen Therapy.
Acronym: OxyFrame
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: OxyFrame
Record Dates: First submitted 2016-03-23; First posted 2016-03-30 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Pulse Oximeter Validation; Long Term Oxygen Therapy; Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy Subjects and patients (Other): Validation of SpO2 sensor in healthy subjects as a first step. Validation of SpO2 sensor in patients as a second step.
  Interventions: Device: OxyFrame

INTERVENTIONS:
Device: OxyFrame — Validation of a miniaturized pulse oximetry sensor for integration into the frame of oxygen delivery glasses.

SUMMARY:
By integrating a miniaturized pulse oximetry sensor into the frame of oxygen delivery glasses which dissimulates the nasal cannula, the investigators hope to optimize and long term oxygen therapy (LTOT) regarding medical and social aspects. The validation of the novel SpO2 sensor is the first step in the concept of personalized, dynamic delivery of oxygen by eyeglasses using a closed-loop system.

DETAILED DESCRIPTION:
Objectives:

1. To determine accuracy of SpO2 measurements by the novel sensor compared to 2 reference pulse oximeters in healthy subjects undergoing a normobaric hypoxic challenge provoking SpO2 desaturation.
2. To determine accuracy of SpO2 measurements by the novel sensor compared to 2 reference pulse oximeters and to arterial blood gas analysis in patients qualifying for LTOT, breathing room air at rest (lying, sitting, standing position) and during exercise (slow walking, 6-MWT, ergometer cycle).

ELIGIBILITY:
Healthy volunteers

Inclusion Criteria:

* Age 18 - 60 years,
* Non smoker,
* Good general health and physical fitness
* Informed Consent

Exclusion Criteria:

* Current or history of tobacco smoking (> 5 py)
* Current alcohol or drug abuse
* Heart disease or untreated arterial hypertension
* Pulmonary disease
* Epilepsy or other major neurologic disease
* Dark skin colour
* Known anemia
* Severe metabolic disease (e.g. diabetes)
* Pregnancy

Patients

Inclusion Criteria:

* Age ≥ 18 years
* Long term oxygen therapy at rest and/or on physical effort
* Hypoxemia in arterial blood gas analysis at rest PaO2 ≤ 55 mmHg or < 60 mmHg with PHT or polycythemia (men Hb > 174 g/L, women Hb > 140 g/L) or:

Oxygen desaturation on effort (SpO2 < 90%)

* Pulmonary disease including Chronic Obstructive Pulmonary Disease, Interstitial Lung Disease and Sarcoidosis
* Informed Consent

Exclusion Criteria:

* Severe hypoxemia (pO2 <40 mmHg)
* Severe hypercapnia (pCO2 >55 mmHg)
* Acute respiratory infection or systemic infection,
* Severe systolic heart disease (LVEF < 25%)
* Myocardial infarction during the last month before inclusion
* Unstable angina pectoris
* Severe aortic stenosis (mean gradient > 40mmHg, valve area <1 cm2)
* Rhythmogenic heart disease
* Severe or untreated arterial hypertension (blood pressure > 180mmHg systolic, >100mmHg diastolic)
* Anemia (Hb < 120 g/l)
* Known or suspected coagulation disorder (e.g. INR > 4)
* Severe or untreated metabolic disorder
* Neurologic disease or dementia
* Pregnancy
* History of non-compliance to medical treatment
* Current alcohol, drug abuse or current tobacco smoking
* Dark skin color

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Assessment of accuracy in patients | At baseline
  Assessment of the accuracy of the novel pulse oximeter sensor in patients qualifying for LTOT over the entire saturation range by calculating accuracy root mean square (ARMS). Continuous SpO2 measurement of the novel pulse oximeter will be compared to measurements assessed by 2 standard pulse oximeters and arterial blood gas analysis.

SECONDARY OUTCOMES:
Assessment of accuracy in healthy volunteers | At baseline
  Assessment of accuracy of the novel pulse oximeter sensor in healthy subjects undergoing a normobaric hypoxic challenge provoking SpO2 desaturation. SpO2 will be measured continuously over the hole procedure and SpO2 range by the novel pulse oximeter sensor and the 2 reference pulse oximeters.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Funke, MD, Principal Investigator — Department of Pulmonary Medicine, University Hospital Bern
Locations (1):
- Department of Pulmonary Medicine, University Hospital Bern, Bern, Canton of Bern, Switzerland